CLINICAL TRIAL: NCT06374329
Title: Effect of Interceptive Strategies on the Clinical Outcome of Impacted Maxillary Permanent Canines - RCT Phase 2
Brief Title: Effect of Interceptive Strategies on the Clinical Outcome of Impacted Maxillary Permanent Canines
Acronym: RCTcanines2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Karolinska Institutet (Other); University of Copenhagen (Other); Palacky University (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S68717
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-04

CONDITIONS: Tooth Impaction; Canine Teeth
MeSH Terms: conditions — Tooth, Impacted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Posterior crossbite and lack of space (Group A - Expansion) (Experimental): Patients with at least one impacted maxillary canine, uni or bilateral posterior crossbite and lack of space in the upper arch will be treated with slow maxillary expansion with removable plates (GROUP A - expansion)
  Interventions: Other: Interceptive Slow Maxillary Expansion with removable plates
- No Posterior crossbite and lack of space (Group B - Expansion) (Experimental): Patients with at least one impacted maxillary canine, no uni or bilateral posterior crossbite and lack of space in the upper arch will be treated with slow maxillary expansion with removable plates (GROUP B - expansion) .
  Inclusion in groups B and C will be randomized
  Interventions: Other: Interceptive Slow Maxillary Expansion with removable plates
- No Posterior crossbite and lack of space (Group C - Expansion) (No Intervention): Patients with at least one impacted maxillary canine, no uni or bilateral posterior crossbite and lack of space in the upper arch will receive no treatment and will be simply followed up (GROUP C - No intervention) Inclusion in groups B and C will be randomized

INTERVENTIONS:
Other: Interceptive Slow Maxillary Expansion with removable plates — Interceptive Slow Maxillary Expansion with removable plates (see Willems et al 2023) https://doi.org/10.1093/ejo/cjad014
  Arms: No Posterior crossbite and lack of space (Group B - Expansion); Posterior crossbite and lack of space (Group A - Expansion)

SUMMARY:
Canine impaction is a sign of abnormal dental development with potentially far-reaching consequences (such as significant root resorption and loss of lateral incisors. This compromises both aesthetics and function of the teeth, making the prediction of canine tooth impaction increasingly important. Interceptive orthodontic measures, such as extraction of deciduous canines or molars or maxillary expansion aim to create extra space in the dental arch, allowing the canines to position themselves better and normalizing their eruption pattern.

This study corresponds to the second phase of an RCT, based on the results of the first phase, published in July 2023 (S59030) (Willems G, Butaye C, Raes M, Zong C, Begnoni G, Cadenas de Llano-Pérula M. Early prevention of maxillary canine impaction: a randomized clinical trial. Eur J Orthod. 31;45(4):359-369). The first phase compared the effect of 3 interceptive strategies (expansion, extraction and no intervention) on the position of impacted maxillary canines, finding that maxillary expansion provides the most improvement on impacted canine position. In second phase, 8-year-old patients without posterior crossbite and lack of space in the dental arch are randomized to treatment with 'slow maxillary expansion with removable plates' or 'no treatment'. These groups are additionally compared with patients with a crossbite and lack of space, which always receive expansion treatment. All selected patients will be followed up for at least 18 months. The primary endpoint is to investigate the effect of maxillary expansion with removable plates on the position of maxillary canines prone to impaction during early mixed dentition, assessed on panoramic X-rays. The secondary endpoint is the assessment of the need for additional orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Female or male patients between 7.5 and 9.5 years-old coming to the department of Orthodontics of UZ Leuven (or one of the participating centres) seeking for orthodontic advice.
* Presenting with one or two impacted maxillary permanent canines, defined by 3¨ML between 15 and 45 degrees (If bilateral impaction occurs, categorization into the different protocol groups will be based on the canine showing the worst position).
* Presenting with one or two maxillary permanent canines showing no more than ¾ root formation, persisting deciduous canines and molars and lack of space in the maxillary arch, defined by ALD>0 mm
* Any race Inclusion criteria Group A: posterior crossbite Inclusion criteria Groups B and C: no posterior crossbite

Exclusion Criteria:

* Fully erupted permanent canines
* Previous orthodontic treatment.
* Canines with completed root formation
* Evidence of root resorption of adjacent teeth or root malformation of the canines that would obligate to extract any adjacent teeth or the canine(s).
* Craniofacial syndromes
* Systemic disease that would impede orthodontic treatment/surgery
* Recent exposure to radiotherapy.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Position of the impacted maxillary canine towards the dental midline (3^ML). | 18 months
  Longitudinal difference in the position of the impacted maxillary canine towards the dental midline (3^ML), measured radiologically on panoramic radiographs before the study and at 18 months follow up

SECONDARY OUTCOMES:
Need for subsequent interventions (extraction of deciduous or permanent teeth, other orthodontic interventions, surgical exposure) | 18 months
  Need for subsequent interventions (extraction of deciduous or permanent teeth, other orthodontic interventions, surgical exposure)

CONTACTS AND LOCATIONS:
Locations (3):
- University Hospitals Leuven - Service of Dentistry, Unit of Orthodontics, Leuven, Belgium
- Institute of Dentistry and Oral Sciences, Faculty of Medicine and Dentistry, Palacký University, Olomouc, Czechia
- Faculty of Dentistry, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Willems G, Butaye C, Raes M, Zong C, Begnoni G, Cadenas de Llano-Perula M. Early prevention of maxillary canine impaction: a randomized clinical trial. Eur J Orthod. 2023 Jul 31;45(4):359-369. doi: 10.1093/ejo/cjad014. PMID 37266982
- See also: Department of Oral Healths Sciences - Orthodontics University KU Leuven, Belgium — http://www.orthodonticsleuven.be/